CLINICAL TRIAL: NCT03799640
Title: Multidirectional Yoga Training to Improve in Healthy Older Participants
Brief Title: Multidirectional Yoga for Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180704
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Standard Yoga; Multi-directional Yoga; Educational Control

STUDY DESIGN:
Intervention Model Description: Comparison of Yoga Interventions
Who Masked: Investigator
Masking Description: Tests will not be performed by the investigators providing the interventions..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Yoga (Experimental): Yoga will be performed using linear forward and backward movements.
  Interventions: Other: Multi-directional Yoga; Other: Educational Control
- Multi-directional Yoga (Experimental): The multidirectional yoga training program will use both simple and complex movement sequences (asana or postures) that include a cognitive component. For example, participants will be taught a movement sequence that includes 16-20 yoga postures that increase in difficulty as the training progresses. .
  Interventions: Other: Standard Yoga; Other: Educational Control
- Educational Control (Experimental): Lectures on Health and Wellness
  Interventions: Other: Standard Yoga; Other: Multi-directional Yoga

INTERVENTIONS:
Other: Standard Yoga — Yoga using standard poses and linear movements
  Arms: Educational Control; Multi-directional Yoga
Other: Multi-directional Yoga — The multidirectional yoga training program will use both simple and complex movement sequences (asana or postures) that include a cognitive component. For example, participants will be taught a movement sequence that includes 16-20 yoga postures that increase in difficulty as the training progresses.
  Arms: Educational Control; Standard Yoga
Other: Educational Control — Lectures on health and fitness
  Arms: Multi-directional Yoga; Standard Yoga

SUMMARY:
Older individuals, 60-90, will be provided regular or cognitively based yoga training. They will then be evaluated using standard cognitive testing devices.

DETAILED DESCRIPTION:
Reductions in executive function are common with age. Along with these declines come reductions in simple functional patterns of daily living such as crossing a street, walking in a crowded area, or performing any functions that occurs in an open (changing) environment. This study will use a newly developed yoga program incorporating multi-directional movements, cognitive challenges and visuomotor disturbances to improve executive function and associated movements in persons over 60 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 60-90 years of age
* Capable of walking 50 feet with or without a walking aid-

Exclusion Criteria:

* Regularly participating in yoga or other balance training program
* Currently participating in another exercise study
* Unable to commit to study duration
* Uncontrolled neuromuscular or cardiovascular disease that prevents participation in an exercise study
* Advised not to exercise by their physician

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox: Picture Sequence Memory Test | 5 minutes
  Measures episodic memory. Participants are asked to reproduce a sequence of pictures that is shown on the screen.
NIH Toolbox Flanker test | 5 minutes
  Measures attention and inhibitory control. Participant focuses on a given stimulus while inhibiting attention to stimuli flanking it.
NIH Toolbox List Sorting test | 5 minutes
  Measures working memory. Participant recalls and sequences different visually and orally presented stimuli.
NIH Toolbox Pattern Comparison Processing Speed test | 5 minutes
  Measures speed of processing. Participants discern whether two side-by-side pictures are the same or not, with 85 seconds to respond to as many items as possible. Items are simple so as to purely measure processing speed.
Walking Executive Function Tests | 10 minutes
  Walking and responding to visual cues presented on a 60 inch monitor.
Timed up-and-go | 5 minutes
  Rising from a chair, circumventing a cone and returning to the chair.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Max Orovitz Laboratories, Coral Gables, Florida
  - Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No